CLINICAL TRIAL: NCT03066596
Title: Promoting Asthma Guidelines and Management Through Technology-Based Intervention and Care Coordination
Acronym: PRAGMATIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-6258; 1R01HL133789 (NIH)
Record Dates: First submitted 2017-02-16; First posted 2017-02-28 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Asthma Childhood

STUDY DESIGN:
Intervention Model Description: Cluster randomized design
Masking Description: Follow up assessments will be collected by blinded interviewers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Multifaceted Prompting Intervention (eMPI) (Experimental): The enhanced MPI program (eMPI) consists of innovative multi-level and team-based strategies to enable providers to effectively and efficiently adopt asthma care guidelines. eMPI uses guideline-based prompts at the time of an office visit to support providers' decision-making, increasing the likelihood that they will recommend corrective actions (i.e., preventive medication prescription) to improve asthma management.
  Interventions: Behavioral: eMPI
- Enhanced Usual Care (eUC) Practices (No Intervention): Participants will receive a review packet of the National Asthma Education and Prevention Program (NAEPP) guidelines and educational resources for families. Children will be assessed for asthma severity and level of control at each visit as part of best-practice care, but active intervention components will not be provided.

INTERVENTIONS:
Behavioral: eMPI — The core elements of the multilevel strategy for implementation include:
  Direct Support for Providers' Delivery of Guideline-Based Care in Practice; Enhancements to Increase the Feasibility and Sustainability of eMPI; Involving Clinic Staff in Promoting and Supporting Use of Guidelines; Building Accountability and Commitment to Guideline-Based Care; Promoting Providers' Understanding, Acceptance, and Use of Guidelines
  Arms: Enhanced Multifaceted Prompting Intervention (eMPI)

SUMMARY:
The overall goal of this research study is to test the effectiveness of a multifaceted and multi-level prompting intervention in a real world urban primary care office setting on improving provider-delivered guideline-based asthma care and reducing asthma morbidity among urban children with persistent or uncontrolled asthma.

DETAILED DESCRIPTION:
Investigators will conduct a cluster randomized trial comparing the intervention to enhanced usual care (eUC) in 20 Bronx practices serving over 5,000 children ages 2-12 years with persistent or uncontrolled asthma. Eleven eUC practices will receive guideline information and assess children's asthma severity and control, but active intervention components will not be provided. Practices will join the study in 4 waves over 4 years (4-6 practices per year). Provider adoption of guidelines and utilization of care in all patients (~5,000) ages 2-12 years with persistent or uncontrolled asthma from intervention and eUC practices will be evaluated using Electronic Health Records (EHR) data and practice-based screening for asthma severity and control. Investigators will also enroll a random subset of 512 caregivers of children with persistent/uncontrolled asthma from both study arms to systematically evaluate caregiver-reported child morbidity outcomes and obtain measures not available in EHR.

Intervention consists of academic detailing in the EHR that follow national asthma guidelines and outreach worker care coordination for patients with persistent or uncontrolled asthma.

Comment: While caregivers reported on child outcomes, caregivers were not subjects of the study. See "Pre-Assignment Details" section within the Participant Flow module for more details.

ELIGIBILITY:
Inclusion Criteria:

The criteria listed below will apply to ~5,000 children from eMPI and eUC practices:

* Physician-diagnosed asthma (based on EHR)
* Persistent or uncontrolled asthma as per clinic assessment. Based on NHLBI guidelines, any one of the following: in past month, > 2 days/week with asthma symptoms, >2 days/week with rescue medication use, >2 days/month with nighttime symptoms, or > 2 episodes in the past year that required systemic corticosteroids
* Age 2 and 12 years, inclusive

Additional inclusion criteria will apply to a subset of 512 of children whose caregivers will be interviewed to obtain caregiver-reported morbidity outcomes:

* Caregiver is able to speak and understand either English or Spanish. Participants unable to read will be eligible as all surveys will be administered verbally by research personnel
* Consent from the primary caregiver, caregiver permission for the child to participate as well as assent from the child (>7 years). If there are eligible siblings, only one child will be randomly selected

Exclusion Criteria:

* The child has other significant medical conditions, such as congenital heart disease, cystic fibrosis, or other chronic lung disease, that could interfere with the assessment of asthma-related measures

Additional exclusion criteria will apply to a subset of 512 children/caregivers as described above:

* No access to a telephone to conduct follow-up surveys
* Children in foster care or other situations in which consent cannot be obtained from a guardian

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 530 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Reznik, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Children's Hospital at Montefiore, Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared for this study. This study predated the 2023 Data Management and Sharing Policy and was subject to the 2003 NIH Data Sharing Policy. Based on this policy it did not meet the requirements for the sharing of research, and therefore IPD, data.

REFERENCES:
- [Background] Bloom B, Jones LI, Freeman G. Summary health statistics for U.S. children: National Health Interview Survey, 2012. Vital Health Stat 10. 2013 Dec;(258):1-81. PMID 24784481
- [Background] Flores G, Snowden-Bridon C, Torres S, Perez R, Walter T, Brotanek J, Lin H, Tomany-Korman S. Urban minority children with asthma: substantial morbidity, compromised quality and access to specialists, and the importance of poverty and specialty care. J Asthma. 2009 May;46(4):392-8. doi: 10.1080/02770900802712971. PMID 19484676
- [Background] Szefler SJ, Mitchell H, Sorkness CA, Gergen PJ, O'Connor GT, Morgan WJ, Kattan M, Pongracic JA, Teach SJ, Bloomberg GR, Eggleston PA, Gruchalla RS, Kercsmar CM, Liu AH, Wildfire JJ, Curry MD, Busse WW. Management of asthma based on exhaled nitric oxide in addition to guideline-based treatment for inner-city adolescents and young adults: a randomised controlled trial. Lancet. 2008 Sep 20;372(9643):1065-72. doi: 10.1016/S0140-6736(08)61448-8. PMID 18805335
- [Background] Wisnivesky JP, Lorenzo J, Lyn-Cook R, Newman T, Aponte A, Kiefer E, Halm EA. Barriers to adherence to asthma management guidelines among inner-city primary care providers. Ann Allergy Asthma Immunol. 2008 Sep;101(3):264-70. doi: 10.1016/S1081-1206(10)60491-7. PMID 18814449
- [Background] Okelo SO, Butz AM, Sharma R, Diette GB, Pitts SI, King TM, Linn ST, Reuben M, Chelladurai Y, Robinson KA. Interventions to modify health care provider adherence to asthma guidelines: a systematic review. Pediatrics. 2013 Sep;132(3):517-34. doi: 10.1542/peds.2013-0779. Epub 2013 Aug 26. PMID 23979092
- [Background] Cabana MD, Rand CS, Powe NR, Wu AW, Wilson MH, Abboud PA, Rubin HR. Why don't physicians follow clinical practice guidelines? A framework for improvement. JAMA. 1999 Oct 20;282(15):1458-65. doi: 10.1001/jama.282.15.1458. PMID 10535437
- [Background] Cabana MD, Ebel BE, Cooper-Patrick L, Powe NR, Rubin HR, Rand CS. Barriers pediatricians face when using asthma practice guidelines. Arch Pediatr Adolesc Med. 2000 Jul;154(7):685-93. doi: 10.1001/archpedi.154.7.685. PMID 10891020
- [Background] Frey SM, Fagnano M, Halterman JS. Caregiver education to promote appropriate use of preventive asthma medications: what is happening in primary care? J Asthma. 2016;53(2):213-9. doi: 10.3109/02770903.2015.1075549. Epub 2015 Aug 18. PMID 26288255
- [Background] Okelo SO, Butz AM, Sharma R, Diette GB, Pitts SI, King TM, Linn ST, Reuben M, Chelladurai Y, Robinson KA. Interventions to Modify Health Care Provider Adherence to Asthma Guidelines [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2013 May. Report No.: 13-EHC022-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK144097/ PMID 23805435
- [Background] Reznik M, Jaramillo Y, Wylie-Rosett J. Demonstrating and assessing metered-dose inhaler-spacer technique: pediatric care providers' self-reported practices and perceived barriers. Clin Pediatr (Phila). 2014 Mar;53(3):270-6. doi: 10.1177/0009922813512521. Epub 2013 Dec 12. PMID 24336438
- [Background] Okelo SO, Siberry GK, Solomon BS, Bilderback AL, Yamazaki M, Hetzler T, Ferrell CL, Dhepyasuwan N, Serwint JR; CORNET Investigators. Asthma treatment decisions by pediatric residents do not consistently conform to guidelines or improve with level of training. Acad Pediatr. 2014 May-Jun;14(3):287-93. doi: 10.1016/j.acap.2013.12.008. Epub 2014 Mar 12. PMID 24629404
- [Background] Shiffman RN, Freudigman Md, Brandt CA, Liaw Y, Navedo DD. A guideline implementation system using handheld computers for office management of asthma: effects on adherence and patient outcomes. Pediatrics. 2000 Apr;105(4 Pt 1):767-73. doi: 10.1542/peds.105.4.767. PMID 10742318
- [Background] Eccles M, McColl E, Steen N, Rousseau N, Grimshaw J, Parkin D, Purves I. Effect of computerised evidence based guidelines on management of asthma and angina in adults in primary care: cluster randomised controlled trial. BMJ. 2002 Oct 26;325(7370):941. doi: 10.1136/bmj.325.7370.941. PMID 12399345
- [Background] Cloutier MM, Hall CB, Wakefield DB, Bailit H. Use of asthma guidelines by primary care providers to reduce hospitalizations and emergency department visits in poor, minority, urban children. J Pediatr. 2005 May;146(5):591-7. doi: 10.1016/j.jpeds.2004.12.017. PMID 15870660
- [Background] Lesho EP, Myers CP, Ott M, Winslow C, Brown JE. Do clinical practice guidelines improve processes or outcomes in primary care? Mil Med. 2005 Mar;170(3):243-6. doi: 10.7205/milmed.170.3.243. PMID 15828703
- [Background] Mitchell EA, Didsbury PB, Kruithof N, Robinson E, Milmine M, Barry M, Newman J. A randomized controlled trial of an asthma clinical pathway for children in general practice. Acta Paediatr. 2005 Feb;94(2):226-33. doi: 10.1111/j.1651-2227.2005.tb01896.x. PMID 15981759
- [Background] Halterman JS, Fisher S, Conn KM, Fagnano M, Lynch K, Marky A, Szilagyi PG. Improved preventive care for asthma: a randomized trial of clinician prompting in pediatric offices. Arch Pediatr Adolesc Med. 2006 Oct;160(10):1018-25. doi: 10.1001/archpedi.160.10.1018. PMID 17018460
- [Background] Martens JD, van der Weijden T, Severens JL, de Clercq PA, de Bruijn DP, Kester AD, Winkens RA. The effect of computer reminders on GPs' prescribing behaviour: a cluster-randomised trial. Int J Med Inform. 2007 Dec;76 Suppl 3:S403-16. doi: 10.1016/j.ijmedinf.2007.04.005. Epub 2007 Jun 14. PMID 17569575
- [Background] Bell LM, Grundmeier R, Localio R, Zorc J, Fiks AG, Zhang X, Stephens TB, Swietlik M, Guevara JP. Electronic health record-based decision support to improve asthma care: a cluster-randomized trial. Pediatrics. 2010 Apr;125(4):e770-7. doi: 10.1542/peds.2009-1385. Epub 2010 Mar 15. PMID 20231191
- [Background] Cho SH, Jeong JW, Park HW, Pyun BY, Chang SI, Moon HB, Kim YY, Choi BW. Effectiveness of a computer-assisted asthma management program on physician adherence to guidelines. J Asthma. 2010 Aug;47(6):680-6. doi: 10.3109/02770903.2010.481342. PMID 20632781
- [Background] Davis AM, Cannon M, Ables AZ, Bendyk H. Using the electronic medical record to improve asthma severity documentation and treatment among family medicine residents. Fam Med. 2010 May;42(5):334-7. PMID 20455109
- [Background] de Vries TW, van den Berg PB, Duiverman EJ, de Jong-van den Berg LT. Effect of a minimal pharmacy intervention on improvement of adherence to asthma guidelines. Arch Dis Child. 2010 Apr;95(4):302-4. doi: 10.1136/adc.2008.145581. Epub 2009 Apr 23. PMID 19395402
- [Background] Ragazzi H, Keller A, Ehrensberger R, Irani AM. Evaluation of a practice-based intervention to improve the management of pediatric asthma. J Urban Health. 2011 Feb;88 Suppl 1(Suppl 1):38-48. doi: 10.1007/s11524-010-9471-3. PMID 21337050
- [Background] Gupta RS, Weiss KB. The 2007 National Asthma Education and Prevention Program asthma guidelines: accelerating their implementation and facilitating their impact on children with asthma. Pediatrics. 2009 Mar;123 Suppl 3:S193-8. doi: 10.1542/peds.2008-2233J. PMID 19221163
- [Background] Shapiro A, Gracy D, Quinones W, Applebaum J, Sarmiento A. Putting guidelines into practice: improving documentation of pediatric asthma management using a decision-making tool. Arch Pediatr Adolesc Med. 2011 May;165(5):412-8. doi: 10.1001/archpediatrics.2011.49. PMID 21536955
- [Background] Wagner EH, Austin BT, Davis C, Hindmarsh M, Schaefer J, Bonomi A. Improving chronic illness care: translating evidence into action. Health Aff (Millwood). 2001 Nov-Dec;20(6):64-78. doi: 10.1377/hlthaff.20.6.64. PMID 11816692
- [Background] Halterman JS, Fagnano M, Tremblay PJ, Fisher SG, Wang H, Rand C, Szilagyi P, Butz A. Prompting asthma intervention in Rochester-uniting parents and providers (PAIR-UP): a randomized trial. JAMA Pediatr. 2014 Oct;168(10):e141983. doi: 10.1001/jamapediatrics.2014.1983. Epub 2014 Oct 6. PMID 25288141
- [Background] Smith LA, Hatcher-Ross JL, Wertheimer R, Kahn RS. Rethinking race/ethnicity, income, and childhood asthma: racial/ethnic disparities concentrated among the very poor. Public Health Rep. 2005 Mar-Apr;120(2):109-16. doi: 10.1177/003335490512000203. PMID 15842111
- [Background] Claudio L, Stingone JA, Godbold J. Prevalence of childhood asthma in urban communities: the impact of ethnicity and income. Ann Epidemiol. 2006 May;16(5):332-40. doi: 10.1016/j.annepidem.2005.06.046. Epub 2005 Oct 20. PMID 16242960
- [Background] Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007. Pediatrics. 2009 Mar;123 Suppl 3:S131-45. doi: 10.1542/peds.2008-2233C. PMID 19221156
- [Background] Bloom B, Cohen RA, Freeman G. Summary health statistics for U.S. children: National Health Interview Survey, 2007. Vital Health Stat 10. 2009 Jan;(239):1-80. PMID 19326838
- [Background] Cabana MD, Lara M, Shannon J. Racial and ethnic disparities in the quality of asthma care. Chest. 2007 Nov;132(5 Suppl):810S-817S. doi: 10.1378/chest.07-1910. PMID 17998345
- [Background] Webber MP, Carpiniello KE, Oruwariye T, Lo Y, Burton WB, Appel DK. Burden of asthma in inner-city elementary schoolchildren: do school-based health centers make a difference? Arch Pediatr Adolesc Med. 2003 Feb;157(2):125-9. doi: 10.1001/archpedi.157.2.125. PMID 12580680
- [Background] Reznik M, Bauman LJ, Okelo SO, Halterman JS. Asthma identification and medication administration forms in New York City schools. Ann Allergy Asthma Immunol. 2015 Jan;114(1):67-68.e1. doi: 10.1016/j.anai.2014.10.006. Epub 2014 Oct 24. No abstract available. PMID 25454012
- [Background] Wu AC, Smith L, Bokhour B, Hohman KH, Lieu TA. Racial/Ethnic variation in parent perceptions of asthma. Ambul Pediatr. 2008 Mar-Apr;8(2):89-97. doi: 10.1016/j.ambp.2007.10.007. PMID 18355737
- [Background] Halterman JS, Auinger P, Conn KM, Lynch K, Yoos HL, Szilagyi PG. Inadequate therapy and poor symptom control among children with asthma: findings from a multistate sample. Ambul Pediatr. 2007 Mar-Apr;7(2):153-9. doi: 10.1016/j.ambp.2006.11.007. PMID 17368410
- [Background] Akinbami LJ, Moorman JE, Simon AE, Schoendorf KC. Trends in racial disparities for asthma outcomes among children 0 to 17 years, 2001-2010. J Allergy Clin Immunol. 2014 Sep;134(3):547-553.e5. doi: 10.1016/j.jaci.2014.05.037. Epub 2014 Aug 1. PMID 25091437
- [Background] Capo-Ramos DE, Duran C, Simon AE, Akinbami LJ, Schoendorf KC. Preventive asthma medication discontinuation among children enrolled in fee-for-service Medicaid. J Asthma. 2014 Aug;51(6):618-26. doi: 10.3109/02770903.2014.895010. Epub 2014 Mar 20. PMID 24580372
- [Background] Cabana MD, Bruckman D, Meister K, Bradley JF, Clark N. Documentation of asthma severity in pediatric outpatient clinics. Clin Pediatr (Phila). 2003 Mar;42(2):121-5. doi: 10.1177/000992280304200204. PMID 12659384
- [Background] Biksey T, Zickmund S, Wu F. Disparities in risk communication: a pilot study of asthmatic children, their parents, and home environments. J Natl Med Assoc. 2011 May;103(5):388-91. doi: 10.1016/s0027-9684(15)30334-5. PMID 21809787
- [Background] Bousquet J, Khaltaev N, Cruz AA, Denburg J, Fokkens WJ, Togias A, Zuberbier T, Baena-Cagnani CE, Canonica GW, van Weel C, Agache I, Ait-Khaled N, Bachert C, Blaiss MS, Bonini S, Boulet LP, Bousquet PJ, Camargos P, Carlsen KH, Chen Y, Custovic A, Dahl R, Demoly P, Douagui H, Durham SR, van Wijk RG, Kalayci O, Kaliner MA, Kim YY, Kowalski ML, Kuna P, Le LT, Lemiere C, Li J, Lockey RF, Mavale-Manuel S, Meltzer EO, Mohammad Y, Mullol J, Naclerio R, O'Hehir RE, Ohta K, Ouedraogo S, Palkonen S, Papadopoulos N, Passalacqua G, Pawankar R, Popov TA, Rabe KF, Rosado-Pinto J, Scadding GK, Simons FE, Toskala E, Valovirta E, van Cauwenberge P, Wang DY, Wickman M, Yawn BP, Yorgancioglu A, Yusuf OM, Zar H, Annesi-Maesano I, Bateman ED, Ben Kheder A, Boakye DA, Bouchard J, Burney P, Busse WW, Chan-Yeung M, Chavannes NH, Chuchalin A, Dolen WK, Emuzyte R, Grouse L, Humbert M, Jackson C, Johnston SL, Keith PK, Kemp JP, Klossek JM, Larenas-Linnemann D, Lipworth B, Malo JL, Marshall GD, Naspitz C, Nekam K, Niggemann B, Nizankowska-Mogilnicka E, Okamoto Y, Orru MP, Potter P, Price D, Stoloff SW, Vandenplas O, Viegi G, Williams D, World Health O, Galen, AllerGen. Allergic Rhinitis and its Impact on Asthma (ARIA) 2008 update (in collaboration with the World Health Organization, GA(2)LEN and AllerGen). Allergy. 2008;63 Suppl 86:8-160.
- [Background] Diaz J, Farzan S. Clinical implications of the obese-asthma phenotypes. Immunol Allergy Clin North Am. 2014 Nov;34(4):739-51. doi: 10.1016/j.iac.2014.07.008. PMID 25282287
- [Background] Scadding G, Walker S. Poor asthma control?--then look up the nose. The importance of co-morbid rhinitis in patients with asthma. Prim Care Respir J. 2012 Jun;21(2):222-8. doi: 10.4104/pcrj.2012.00035. PMID 22643359
- [Background] Lee MG, Cross KJ, Yang WY, Sutton BS, Jiroutek MR. Frequency of asthma education in primary care in the years 2007-2010. J Asthma. 2016;53(2):220-6. doi: 10.3109/02770903.2015.1087024. Epub 2015 Sep 18. PMID 26313596
- [Background] McMullen A, Yoos HL, Anson E, Kitzmann H, Halterman JS, Arcoleo KS. Asthma care of children in clinical practice: do parents report receiving appropriate education? Pediatr Nurs. 2007 Jan-Feb;33(1):37-44. PMID 17410999
- [Background] Reznik M, Silver EJ, Cao Y. Evaluation of MDI-spacer utilization and technique in caregivers of urban minority children with persistent asthma. J Asthma. 2014 Mar;51(2):149-54. doi: 10.3109/02770903.2013.854379. Epub 2013 Oct 22. PMID 24131031
- [Background] Conn KM, Halterman JS, Lynch K, Cabana MD. The impact of parents' medication beliefs on asthma management. Pediatrics. 2007 Sep;120(3):e521-6. doi: 10.1542/peds.2006-3023. PMID 17766496
- [Background] Mitchell SJ, Bilderback AL, Okelo SO. Racial Disparities in Asthma Morbidity Among Pediatric Patients Seeking Asthma Specialist Care. Acad Pediatr. 2016 Jan-Feb;16(1):64-7. doi: 10.1016/j.acap.2015.06.010. Epub 2015 Aug 29. PMID 26329015
- [Background] James CV, Rosenbaum S. Paying for quality care: implications for racial and ethnic health disparities in pediatric asthma. Pediatrics. 2009 Mar;123 Suppl 3:S205-10. doi: 10.1542/peds.2008-2233L. PMID 19221165
- [Background] Tsuyuki RT, Sin DD, Sharpe HM, Cowie RL, Nilsson C, Man SF; Alberta Strategy to Help Manage Asthma (ASTHMA) Investigators. Management of asthma among community-based primary care physicians. J Asthma. 2005 Apr;42(3):163-7. PMID 15962871
- [Background] Powell BJ, Waltz TJ, Chinman MJ, Damschroder LJ, Smith JL, Matthieu MM, Proctor EK, Kirchner JE. A refined compilation of implementation strategies: results from the Expert Recommendations for Implementing Change (ERIC) project. Implement Sci. 2015 Feb 12;10:21. doi: 10.1186/s13012-015-0209-1. PMID 25889199
- [Background] Butz AM, Walker J, Land CL, Vibbert C, Winkelstein M. Improving asthma communication in high-risk children. J Asthma. 2007 Nov;44(9):739-45. doi: 10.1080/02770900701595683. PMID 17994404
- [Background] Kattan M, Crain EF, Steinbach S, Visness CM, Walter M, Stout JW, Evans R 3rd, Smartt E, Gruchalla RS, Morgan WJ, O'Connor GT, Mitchell HE. A randomized clinical trial of clinician feedback to improve quality of care for inner-city children with asthma. Pediatrics. 2006 Jun;117(6):e1095-103. doi: 10.1542/peds.2005-2160. PMID 16740812
- [Background] Vernacchio L, Francis ME, Epstein DM, Santangelo J, Trudell EK, Reynolds ME, Risko W. Effectiveness of an asthma quality improvement program designed for maintenance of certification. Pediatrics. 2014 Jul;134(1):e242-8. doi: 10.1542/peds.2013-2643. Epub 2014 Jun 16. PMID 24935994
- [Background] Richman MJ, Poltawsky JS. Partnership for excellence in asthma care: evidence-based disease management. Stud Health Technol Inform. 2000;76:107-21. PMID 10947496
- [Background] Baker R, Fraser RC, Stone M, Lambert P, Stevenson K, Shiels C. Randomised controlled trial of the impact of guidelines, prioritized review criteria and feedback on implementation of recommendations for angina and asthma. Br J Gen Pract. 2003 Apr;53(489):284-91. PMID 12879828
- [Background] Coleman CI, Reddy P, Laster-Bradley NM, Dorval S, Munagala B, White CM. Effect of practitioner education on adherence to asthma treatment guidelines. Ann Pharmacother. 2003 Jul-Aug;37(7-8):956-61. doi: 10.1345/aph.1C506. PMID 12841800
- [Background] Schneider A, Wensing M, Biessecker K, Quinzler R, Kaufmann-Kolle P, Szecsenyi J. Impact of quality circles for improvement of asthma care: results of a randomized controlled trial. J Eval Clin Pract. 2008 Apr;14(2):185-90. doi: 10.1111/j.1365-2753.2007.00827.x. Epub 2007 Dec 13. PMID 18093108
- [Background] Daniels EC, Bacon J, Denisio S, Fry YW, Murray V, Quarshie A, Rust G. Translation squared: improving asthma care for high-disparity populations through a safety net practice-based research network. J Asthma. 2005 Jul-Aug;42(6):499-505. doi: 10.1081/JAS-67598. PMID 16293546
- [Background] Frankowski BL, Keating K, Rexroad A, Delaney T, McEwing SM, Wasko N, Lynn S, Shaw J. Community collaboration: concurrent physician and school nurse education and cooperation increases the use of asthma action plans. J Sch Health. 2006 Aug;76(6):303-6. doi: 10.1111/j.1746-1561.2006.00117.x. No abstract available. PMID 16918860
- [Background] Yawn BP, Bertram S, Wollan P. Introduction of Asthma APGAR tools improve asthma management in primary care practices. J Asthma Allergy. 2008 Aug 31;1:1-10. doi: 10.2147/jaa.s3595. PMID 21436980
- [Background] Bender BG, Dickinson P, Rankin A, Wamboldt FS, Zittleman L, Westfall JM. The Colorado Asthma Toolkit Program: a practice coaching intervention from the High Plains Research Network. J Am Board Fam Med. 2011 May-Jun;24(3):240-8. doi: 10.3122/jabfm.2011.03.100171. PMID 21551395
- [Background] Lob SH, Boer JH, Porter PG, Nunez D, Fox P. Promoting best-care practices in childhood asthma: quality improvement in community health centers. Pediatrics. 2011 Jul;128(1):20-8. doi: 10.1542/peds.2010-1962. Epub 2011 Jun 13. PMID 21669890
- [Background] Evans D, Sheares BJ, Vazquez TL. Educating health professionals to improve quality of care for asthma. Paediatr Respir Rev. 2004 Dec;5(4):304-10. doi: 10.1016/j.prrv.2004.07.007. PMID 15531255
- [Background] Lozano P, Finkelstein JA, Carey VJ, Wagner EH, Inui TS, Fuhlbrigge AL, Soumerai SB, Sullivan SD, Weiss ST, Weiss KB. A multisite randomized trial of the effects of physician education and organizational change in chronic-asthma care: health outcomes of the Pediatric Asthma Care Patient Outcomes Research Team II Study. Arch Pediatr Adolesc Med. 2004 Sep;158(9):875-83. doi: 10.1001/archpedi.158.9.875. PMID 15351753
- [Background] Glasgow RE, Nutting PA, King DK, Nelson CC, Cutter G, Gaglio B, Rahm AK, Whitesides H, Amthauer H. A practical randomized trial to improve diabetes care. J Gen Intern Med. 2004 Dec;19(12):1167-74. doi: 10.1111/j.1525-1497.2004.30425.x. PMID 15610326
- [Background] Tunis SR, Stryer DB, Clancy CM. Practical clinical trials: increasing the value of clinical research for decision making in clinical and health policy. JAMA. 2003 Sep 24;290(12):1624-32. doi: 10.1001/jama.290.12.1624. PMID 14506122
- [Background] Institute of Medicine (US) Committee on Understanding and Eliminating Racial and Ethnic Disparities in Health Care; Smedley BD, Stith AY, Nelson AR, editors. Unequal Treatment: Confronting Racial and Ethnic Disparities in Health Care. Washington (DC): National Academies Press (US); 2003. Available from http://www.ncbi.nlm.nih.gov/books/NBK220358/ PMID 25032386
- [Background] Mason T, Wilkinson GW, Nannini A, Martin CM, Fox DJ, Hirsch G. Winning policy change to promote community health workers: lessons from massachusetts in the health reform era. Am J Public Health. 2011 Dec;101(12):2211-6. doi: 10.2105/AJPH.2011.300402. Epub 2011 Oct 20. PMID 22021281
- [Background] Margellos-Anast H, Gutierrez MA, Whitman S. Improving asthma management among African-American children via a community health worker model: findings from a Chicago-based pilot intervention. J Asthma. 2012 May;49(4):380-9. doi: 10.3109/02770903.2012.660295. Epub 2012 Feb 21. PMID 22348448
- [Background] Campbell JD, Brooks M, Hosokawa P, Robinson J, Song L, Krieger J. Community Health Worker Home Visits for Medicaid-Enrolled Children With Asthma: Effects on Asthma Outcomes and Costs. Am J Public Health. 2015 Nov;105(11):2366-72. doi: 10.2105/AJPH.2015.302685. Epub 2015 Aug 13. PMID 26270287
- [Background] Reznik M, Silver EJ, Jaramillo Y. A Randomized Trial of a Community Health Worker (CHW) Led Asthma Intervention: Preliminary Findings. 2014 Pediatric Academic Societies and Asian Society for Pediatric Research Joint Meeting, Vancouver, BC, Canada May 3-6, 2014.
- [Background] Peretz PJ, Matiz LA, Findley S, Lizardo M, Evans D, McCord M. Community health workers as drivers of a successful community-based disease management initiative. Am J Public Health. 2012 Aug;102(8):1443-6. doi: 10.2105/AJPH.2011.300585. Epub 2012 Apr 19. PMID 22515859
- [Background] Fisher-Owens SA, Boddupalli G, Thyne SM. Telephone case management for asthma: an acceptable and effective intervention within a diverse pediatric population. J Asthma. 2011 Mar;48(2):156-61. doi: 10.3109/02770903.2011.554938. PMID 21332378
- [Background] Garbutt JM, Sylvia S, Rook S, Schmandt M, Ruby-Ziegler C, Luby J, Strunk RC. Peer training to improve parenting and childhood asthma management skills: a pilot study. Ann Allergy Asthma Immunol. 2015 Feb;114(2):148-9. doi: 10.1016/j.anai.2014.10.023. Epub 2014 Dec 15. No abstract available. PMID 25524747
- [Background] Garbutt JM, Yan Y, Highstein G, Strunk RC. A cluster-randomized trial shows telephone peer coaching for parents reduces children's asthma morbidity. J Allergy Clin Immunol. 2015 May;135(5):1163-70.e1-2. doi: 10.1016/j.jaci.2014.09.033. Epub 2014 Oct 30. PMID 25445827
- [Background] Thorpe KE, Zwarenstein M, Oxman AD, Treweek S, Furberg CD, Altman DG, Tunis S, Bergel E, Harvey I, Magid DJ, Chalkidou K. A pragmatic-explanatory continuum indicator summary (PRECIS): a tool to help trial designers. CMAJ. 2009 May 12;180(10):E47-57. doi: 10.1503/cmaj.090523. Epub 2009 Apr 16. No abstract available. PMID 19372436
- [Background] Rapkin BD, Weiss ES, Lounsbury DW, Thompson HS, Goodman RM, Schechter CB, Merzel C, Shelton RC, Blank AE, Erb-Downward J, Williams A, Valera P, Padgett DK. Using the interactive systems framework to support a quality improvement approach to dissemination of evidence-based strategies to promote early detection of breast cancer: planning a comprehensive dynamic trial. Am J Community Psychol. 2012 Dec;50(3-4):497-517. doi: 10.1007/s10464-012-9518-6. PMID 22618023
- [Background] Rapkin B.D., Trickett E.J. Comprehensive Dynamic Trial Designs for Behavioral Prevention Research with Communities: Overcoming Inadequacies of the Randomized Controlled Trial Paradigm. In Community Interventions and AIDS. Eds. Trickett E.J. and Pequegnat W. Oxford University Press. 2005:249-277University Press. 2005:249-277.
- [Background] Reznik M, Bauman LJ. Barriers to Physical Activity in Schoolchildren with Asthma: A Parent Perspective Clinical and Translational Science 2012;5(2):168.
- [Background] Brown JV, Bakeman R, Celano MP, Demi AS, Kobrynski L, Wilson SR. Home-based asthma education of young low-income children and their families. J Pediatr Psychol. 2002 Dec;27(8):677-88. doi: 10.1093/jpepsy/27.8.677. PMID 12403858
- [Background] Reznik M, Wylie-Rosett J, Kim M, Ozuah PO. A classroom-based physical activity intervention for urban kindergarten and first-grade students: a feasibility study. Child Obes. 2015 Jun;11(3):314-24. doi: 10.1089/chi.2014.0090. Epub 2015 Mar 6. PMID 25747719
- [Background] Halterman JS, Riekert K, Bayer A, Fagnano M, Tremblay P, Blaakman S, Borrelli B. A pilot study to enhance preventive asthma care among urban adolescents with asthma. J Asthma. 2011 Jun;48(5):523-30. doi: 10.3109/02770903.2011.576741. PMID 21599562
- [Background] Halterman JS, Szilagyi PG, Fisher SG, Fagnano M, Tremblay P, Conn KM, Wang H, Borrelli B. Randomized controlled trial to improve care for urban children with asthma: results of the School-Based Asthma Therapy trial. Arch Pediatr Adolesc Med. 2011 Mar;165(3):262-8. doi: 10.1001/archpediatrics.2011.1. PMID 21383275
- [Background] Rinke ML, Chen AR, Bundy DG, Colantuoni E, Fratino L, Drucis KM, Panton SY, Kokoszka M, Budd AP, Milstone AM, Miller MR. Implementation of a central line maintenance care bundle in hospitalized pediatric oncology patients. Pediatrics. 2012 Oct;130(4):e996-e1004. doi: 10.1542/peds.2012-0295. Epub 2012 Sep 3. PMID 22945408
- [Background] Rinke ML, Dietrich E, Kodeck T, Westcoat K. Operation care: a pilot case management intervention for frequent emergency medical system users. Am J Emerg Med. 2012 Feb;30(2):352-7. doi: 10.1016/j.ajem.2010.12.012. Epub 2011 Jan 26. PMID 21269790
- [Background] Basu Roy U, Michel T, Carpenter A, Lounsbury DW, Sabino E, Stevenson AJ, Combs S, Jacobs J, Padgett D, Rapkin BD. Community-led cancer action councils in Queens, New York: process evaluation of an innovative partnership with the Queens library system. Prev Chronic Dis. 2014 Feb 6;11:130176. doi: 10.5888/pcd11.130176. PMID 24503342
- [Background] Blaakman S, Tremblay PJ, Halterman JS, Fagnano M, Borrelli B. Implementation of a community-based secondhand smoke reduction intervention for caregivers of urban children with asthma: process evaluation, successes and challenges. Health Educ Res. 2013 Feb;28(1):141-52. doi: 10.1093/her/cys070. Epub 2012 Jun 20. PMID 22717938
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Wagner EH. Chronic disease management: what will it take to improve care for chronic illness? Eff Clin Pract. 1998 Aug-Sep;1(1):2-4. No abstract available. PMID 10345255
- [Background] Ockene JK, Zapka JG. Provider education to promote implementation of clinical practice guidelines. Chest. 2000 Aug;118(2 Suppl):33S-39S. doi: 10.1378/chest.118.2_suppl.33s. PMID 10939997
- [Background] Soumerai SB, Avorn J. Principles of educational outreach ('academic detailing') to improve clinical decision making. JAMA. 1990 Jan 26;263(4):549-56. PMID 2104640
- [Background] Halterman JS, McConnochie KM, Conn KM, Yoos HL, Callahan PM, Neely TL, Szilagyi PG. A randomized trial of primary care provider prompting to enhance preventive asthma therapy. Arch Pediatr Adolesc Med. 2005 May;159(5):422-7. doi: 10.1001/archpedi.159.5.422. PMID 15867114
- [Background] Cabana MD, Slish KK, Evans D, Mellins RB, Brown RW, Lin X, Kaciroti N, Clark NM. Impact of Physician Asthma Care Education on patient outcomes. Health Educ Behav. 2014 Oct;41(5):509-17. doi: 10.1177/1090198114547510. PMID 25270176
- [Background] Allen FC, Vargas PA, Kolodner K, Eggleston P, Butz A, Huss K, Malveaux F, Rand CS. Assessing pediatric clinical asthma practices and perceptions: a new instrument. J Asthma. 2000 Feb;37(1):31-42. doi: 10.3109/02770900009055426. PMID 10724296
- [Background] Cabana MD, Slish KK, Evans D, Mellins RB, Brown RW, Lin X, Kaciroti N, Clark NM. Impact of physician asthma care education on patient outcomes. Pediatrics. 2006 Jun;117(6):2149-57. doi: 10.1542/peds.2005-1055. PMID 16740859
- [Background] Clark NM, Gong M, Schork MA, Maiman LA, Evans D, Hurwitz ME, Roloff D, Mellins RB. A scale for Assessing Health Care Providers' Teaching and Communication Behavior regarding asthma. Health Educ Behav. 1997 Apr;24(2):245-56. doi: 10.1177/109019819702400211. PMID 9079582
- [Background] Reddel HK, Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, Casale TB, Chanez P, Enright PL, Gibson PG, de Jongste JC, Kerstjens HA, Lazarus SC, Levy ML, O'Byrne PM, Partridge MR, Pavord ID, Sears MR, Sterk PJ, Stoloff SW, Sullivan SD, Szefler SJ, Thomas MD, Wenzel SE; American Thoracic Society/European Respiratory Society Task Force on Asthma Control and Exacerbations. An official American Thoracic Society/European Respiratory Society statement: asthma control and exacerbations: standardizing endpoints for clinical asthma trials and clinical practice. Am J Respir Crit Care Med. 2009 Jul 1;180(1):59-99. doi: 10.1164/rccm.200801-060ST. PMID 19535666
- [Background] Busse WW, Morgan WJ, Taggart V, Togias A. Asthma outcomes workshop: overview. J Allergy Clin Immunol. 2012 Mar;129(3 Suppl):S1-8. doi: 10.1016/j.jaci.2011.12.985. PMID 22386504
- [Background] Schatz M, Zeiger RS, Drane A, Harden K, Cibildak A, Oosterman JE, Kosinski M. Reliability and predictive validity of the Asthma Control Test administered by telephone calls using speech recognition technology. J Allergy Clin Immunol. 2007 Feb;119(2):336-43. doi: 10.1016/j.jaci.2006.08.042. Epub 2006 Dec 27. PMID 17194469
- [Background] Juniper EF, Guyatt GH, Feeny DH, Ferrie PJ, Griffith LE, Townsend M. Measuring quality of life in the parents of children with asthma. Qual Life Res. 1996 Feb;5(1):27-34. doi: 10.1007/BF00435966. PMID 8901364
- [Background] Asmussen L, Olson LM, Grant EN, Fagan J, Weiss KB. Reliability and validity of the Children's Health Survey for Asthma. Pediatrics. 1999 Dec;104(6):e71. doi: 10.1542/peds.104.6.e71. PMID 10586005
- [Background] Horne R WJ HM. The beliefs about medicines questionnaire: The development and evaluation of a new method for assessing the cognitive representation of medication. Psych Health. 1999.
- [Background] Pak L, Allen PJ. The impact of maternal depression on children with asthma. Pediatr Nurs. 2012 Jan-Feb;38(1):11-9, 30. PMID 22474854
- [Background] Otsuki M, Eakin MN, Arceneaux LL, Rand CS, Butz AM, Riekert KA. Prospective relationship between maternal depressive symptoms and asthma morbidity among inner-city African American children. J Pediatr Psychol. 2010 Aug;35(7):758-67. doi: 10.1093/jpepsy/jsp091. Epub 2009 Oct 22. PMID 19850709
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Clark NM, Gong M, Schork MA, Evans D, Roloff D, Hurwitz M, Maiman L, Mellins RB. Impact of education for physicians on patient outcomes. Pediatrics. 1998 May;101(5):831-6. doi: 10.1542/peds.101.5.831. PMID 9565410
- [Background] Maly RC, Leake B, Silliman RA. Breast cancer treatment in older women: impact of the patient-physician interaction. J Am Geriatr Soc. 2004 Jul;52(7):1138-45. doi: 10.1111/j.1532-5415.2004.52312.x. PMID 15209652
- [Background] Maly RC, Leake B, Silliman RA. Health care disparities in older patients with breast carcinoma: informational support from physicians. Cancer. 2003 Mar 15;97(6):1517-27. doi: 10.1002/cncr.11211. PMID 12627517
- [Background] Maly RC, Frank JC, Marshall GN, DiMatteo MR, Reuben DB. Perceived efficacy in patient-physician interactions (PEPPI): validation of an instrument in older persons. J Am Geriatr Soc. 1998 Jul;46(7):889-94. doi: 10.1111/j.1532-5415.1998.tb02725.x. PMID 9670878
- [Background] MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. Psychol Methods. 2002 Mar;7(1):83-104. doi: 10.1037/1082-989x.7.1.83. PMID 11928892
- [Background] Imai K, Keele L, Tingley D. A general approach to causal mediation analysis. Psychol Methods. 2010 Dec;15(4):309-34. doi: 10.1037/a0020761. PMID 20954780
- [Background] Imai K, Keele L, Tingley D, Yamamoto T (2010). Causal Mediation Analysis Using R.
- [Background] Rubin, D.B. (1976) Inference and missing data. Biometrika, 63, 581-592.
- [Background] Finkelstein JA, Lozano P, Streiff KA, Arduino KE, Sisk CA, Wagner EH, Weiss KB, Inui TS. Clinical effectiveness research in managed-care systems: lessons from the Pediatric Asthma Care PORT. Patient Outcomes Research Team. Health Serv Res. 2002 Jun;37(3):775-89. doi: 10.1111/1475-6773.00048. PMID 12132605
- [Background] Fuhlbrigge AL, Kitch BT, Paltiel AD, Kuntz KM, Neumann PJ, Dockery DW, Weiss ST. FEV(1) is associated with risk of asthma attacks in a pediatric population. J Allergy Clin Immunol. 2001 Jan;107(1):61-7. doi: 10.1067/mai.2001.111590. PMID 11149992
- [Background] Jenkins HA, Cherniack R, Szefler SJ, Covar R, Gelfand EW, Spahn JD. A comparison of the clinical characteristics of children and adults with severe asthma. Chest. 2003 Oct;124(4):1318-24. doi: 10.1378/chest.124.4.1318. PMID 14555561
- [Background] Sharek PJ, Mayer ML, Loewy L, Robinson TN, Shames RS, Umetsu DT, Bergman DA. Agreement among measures of asthma status: a prospective study of low-income children with moderate to severe asthma. Pediatrics. 2002 Oct;110(4):797-804. doi: 10.1542/peds.110.4.797. PMID 12359798
- [Background] Bacharier LB MD, Lemanske RF, Schend V, Sorkness C, Strunk RC. Classifying asthma severity in children: is measuring lung function helpful? . J Allergy Clin Immunol. 2002.
- [Background] Spahn JD, Cherniack R, Paull K, Gelfand EW. Is forced expiratory volume in one second the best measure of severity in childhood asthma? Am J Respir Crit Care Med. 2004 Apr 1;169(7):784-6. doi: 10.1164/rccm.200309-1234OE. Epub 2004 Jan 30. No abstract available. PMID 14754761
- [Result] Reznik M, Ball-Jones R, Ibarra J. The COVID-19 pandemic and asthma management: a family caregiver perspective. J Asthma. 2025 May;62(5):817-823. doi: 10.1080/02770903.2024.2447285. Epub 2025 Jan 8. PMID 39726143
- [Result] Telzak A, Fiori KP, Chambers EC, Haughton J, Levano S, Reznik M. Unmet Social Needs and Pediatric Asthma Severity in an Urban Primary Care Setting. Acad Pediatr. 2023 Sep-Oct;23(7):1361-1367. doi: 10.1016/j.acap.2023.02.009. Epub 2023 Feb 27. PMID 36858248
- See also: National Heart Lung and Blood Institute. National Asthma Education and Prevention Program. Expert panel report 3: guidelines for the diagnosis and management of asthma. NIH Publication Number 08 5846. Bethesda, MD: 2007. — http://www.nhlbi.nih.gov/guidelines/asthma/
- See also: Patient-Centered Medical Home Recognition. — http://www.ncqa.org/Programs/Recognition/Practices/PatientCenteredMedicalHomePCMH.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Because children with asthma (ages 2-12) were the subjects of the study, caregivers had to complete validated surveys/questionnaires in order to collect child-specific data and outcome measures about their child's asthma. The study was exclusively for children with asthma. Parents were not subjects in the study.
Units Other Than Participants: clinic
Groups:
- Enhanced Multifaceted Prompting Intervention (eMPI): The enhanced MPI program (eMPI) consists of innovative multi-level and team-based strategies to enable providers to effectively and efficiently adopt asthma care guidelines. eMPI uses guideline-based prompts at the time of an office visit to support providers' decision-making, increasing the likelihood that they will recommend corrective actions (i.e., preventive medication prescription) to improve asthma management.
  eMPI: The core elements of the multilevel strategy for implementation include:
  Direct Support for Providers' Delivery of Guideline-Based Care in Practice; Enhancements to Increase the Feasibility and Sustainability of eMPI; Involving Clinic Staff in Promoting and Supporting Use of Guidelines; Building Accountability and Commitment to Guideline-Based Care; Promoting Providers' Understanding, Acceptance, and Use of Guidelines
Period: Overall Study
Arm/Group | Enhanced Multifaceted Prompting Intervention (eMPI) | Enhanced Usual Care (eUC) Practices
Started | 265; 9 clinic | 265; 9 clinic
Completed | 247; 9 clinic | 253; 9 clinic
Not Completed | 18; 0 clinic | 12; 0 clinic
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 14 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Multifaceted Prompting Intervention (eMPI) | Enhanced Usual Care (eUC) Practices | Total
Number analyzed (Participants) | 265 | 265 | 530
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.65 (2.75) | 6.68 (2.94) | 6.66 (2.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 95 | 204
  Male | 156 | 170 | 326
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 184 | 180 | 364
  Not Hispanic or Latino | 79 | 84 | 163
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 103 | 107 | 210
  White | 30 | 23 | 53
  More than one race | 46 | 56 | 102
  Unknown or Not Reported | 82 | 75 | 157
Region of Enrollment [Number; unit: participants]
  United States | 265 | 265 | 530

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 1 or More Guideline-based Corrective Actions Taken
Description: The percentage of participants with 1 or more guideline-based corrective actions taken (i.e., controller medication prescription or adjustment, trigger evaluation), as recorded in the electronic health record (EHR) is reported. Results are summarized in number/percentage of participants with 1 or more guideline-based corrective actions taken by study arm.
Time Frame: Immediately post-intervention, up to 1 year
Population: All randomized subjects were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Multifaceted Prompting Intervention (eMPI) | Enhanced Usual Care (eUC) Practices
Number analyzed (Participants) | 265 | 265
Participants | 241 | 197
Statistical Analysis 1: Comparison: Enhanced Multifaceted Prompting Intervention (eMPI) vs Enhanced Usual Care (eUC) Practices; Test type: Superiority — A generalized linear model (GLM) with logit link function was used to compare the percentage of participants with corrected actions taken and GEE method was used to account for within-clinic correlation. The null hypothesis is that there is no difference between groups in the the percentage of participants with corrected actions taken. With 530 participants at baseline, ≤10% attrition at 12 months, the study has greater than 80% power to detect a difference of 15 percentage points; p < .001, GLM with GEE — The p-values reported above represented the calculated value rather than predetermined thresholds for significance. Statistical significance was defined as a p-value less than 0.05; Odds Ratio (OR) = 3.47, 95% CI 2-sided [1.98 to 6.08]
Statistical Analysis 2: Comparison: Enhanced Multifaceted Prompting Intervention (eMPI) vs Enhanced Usual Care (eUC) Practices; Test type: Superiority — This analysis is similar to analysis 1, however, the model adjusting for sex, age, race/ethnicity, symptom free days (at baseline), nurse screening results, clinic characteristics, visit type, caregiver education, and smoking exposure (at baseline); p < .001, GLM with GEE — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.66, 95% CI 2-sided [1.97 to 6.82]

2. Secondary Outcome: Symptom Free Days (SFDs)
Description: The number of days without symptoms during the past 14 days is summarized by study arm at baseline and every 3 months up through the 12 month follow up evaluation.
Time Frame: Baseline, and 3 month, 6 month, 9 month, and 12 month follow-up evaluations
Population: The number of participants analyzed at each timepoint for both arms is depicted in the table below.
Measure: Mean (Standard Deviation); unit: number of symptom free days
Arm/Group | Enhanced Multifaceted Prompting Intervention (eMPI) | Enhanced Usual Care (eUC) Practices
Number analyzed (Participants) | 265 | 265
number of symptom free days
  Baseline | 5.79 (4.70) | 6.41 (4.72)
  3 month: number analyzed (Participants) | 253 | 255
  3 month | 9.33 (4.95) | 9.17 (4.82)
  6 month: number analyzed (Participants) | 250 | 250
  6 month | 9.68 (4.52) | 10.33 (4.06)
  9 month: number analyzed (Participants) | 244 | 241
  9 month | 10.07 (4.37) | 10.78 (4.36)
  12 month: number analyzed (Participants) | 247 | 253
  12 month | 10.53 (4.16) | 10.44 (4.49)
Statistical Analysis 1: Comparison: Enhanced Multifaceted Prompting Intervention (eMPI) vs Enhanced Usual Care (eUC) Practices; 3 month follow up; Test type: Superiority — A generalized linear model (GLM) with generalized estimating equations (GEE) was used to compare changes over time between the two groups in symptom-free days (SFDs) during the past two weeks, accounting for within-subject correlation. The null hypothesis at each time point was that there is no difference between groups in the change in SFDs. With 530 participants at baseline, ≤10% attrition at 12 months, the study has 80% power to detect a standardized effect size >0.29; p = 0.174, GLM with GEE; Ratio of Rate Ratios = 1.13, 95% CI 2-sided [0.95 to 1.34]
Statistical Analysis 2: Comparison: Enhanced Multifaceted Prompting Intervention (eMPI) vs Enhanced Usual Care (eUC) Practices; 6 month follow up; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.741, GLM with GEE; Ratio of Rate Ratios = 1.04, 95% CI 2-sided [0.85 to 1.27]
Statistical Analysis 3: Comparison: Enhanced Multifaceted Prompting Intervention (eMPI) vs Enhanced Usual Care (eUC) Practices; 9 month follow up; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.724, GLM with GEE; Ratio of Rate Ratios = 1.03, 95% CI 2-sided [0.85 to 1.25]
Statistical Analysis 4: Comparison: Enhanced Multifaceted Prompting Intervention (eMPI) vs Enhanced Usual Care (eUC) Practices; 12 month follow up; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.229, GLM with GEE; Ratio of Rate Ratios = 1.12, 95% CI 2-sided [0.93 to 1.34]
Statistical Analysis 5: Comparison: Enhanced Multifaceted Prompting Intervention (eMPI) vs Enhanced Usual Care (eUC) Practices; 3 month follow up; Test type: Superiority — This analysis is similar to Analysis 1, with adjustment for baseline outcome (symptom-free days) and seasonality; p = 0.186, GLM with GEE; Ratio of Rate Ratios = 1.13, 95% CI 2-sided [0.94 to 1.34]
Statistical Analysis 6: Comparison: Enhanced Multifaceted Prompting Intervention (eMPI) vs Enhanced Usual Care (eUC) Practices; 6 month follow up; Test type: Superiority — This analysis is similar to Analysis 2, with adjustment for baseline outcome (symptom-free days) and seasonality; p = 0.744, GLM with GEE; Ratio of Rate Ratios = 1.04, 95% CI 2-sided [0.84 to 1.27]
Statistical Analysis 7: Comparison: Enhanced Multifaceted Prompting Intervention (eMPI) vs Enhanced Usual Care (eUC) Practices; 9 month follow up; Test type: Superiority — This analysis is similar to Analysis 3, with adjustment for baseline outcome (symptom-free days) and seasonality; p = 0.765, GLM with GEE; Ratio of Rate Ratios = 1.03, 95% CI 2-sided [0.85 to 1.25]
Statistical Analysis 8: Comparison: Enhanced Multifaceted Prompting Intervention (eMPI) vs Enhanced Usual Care (eUC) Practices; 12 month follow up; Test type: Superiority — This analysis is similar to Analysis 4, with adjustment for baseline outcome (symptom-free days) and seasonality; p = 0.241, GLM with GEE; Ratio of Rate Ratios = 1.11, 95% CI 2-sided [0.93 to 1.33]

3. Other Pre Specified Outcome: Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ)
Description: caregiver asthma related quality of life
Time Frame: every 3 months up to 12 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Health Care Utilization: Number of ED Visits for Asthma
Description: number of ED visits for asthma
Time Frame: every 3 months up to 12 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Health Care Utilization: Number Hospitalizations for Asthma
Description: number hospitalizations for asthma
Time Frame: every 3 months up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Enhanced Multifaceted Prompting Intervention (eMPI) | Enhanced Usual Care (eUC) Practices
All-Cause Mortality (participants affected / at risk) | 0/265 | 0/265
Serious Adverse Events (participants affected / at risk) | 0/265 | 0/265
Other Adverse Events (participants affected / at risk) | 0/265 | 0/265

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT03066596/Prot_SAP_000.pdf